CLINICAL TRIAL: NCT02503501
Title: A Phase II, Single Center, Randomized, Double-Blind, Placebo-Controlled Study of the Safety and the Therapeutic Effectiveness of Intranasal Glulisine in Amnestic Mild Cognitive Impairment and Probable Mild Alzheimer's Disease
Brief Title: Intranasal Glulisine in Amnestic Mild Cognitive Impairment and Probable Mild Alzheimer's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study will not have power to show a difference between groups.
Sponsor: HealthPartners Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IN-INSUL-MCI-AD
Record Dates: First submitted 2015-07-14; First posted 2015-07-21 (Estimated); Results first posted 2020-04-09 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-01

CONDITIONS: Mild Cognitive Impairment; Alzheimer's Disease (AD)
Keywords: Memory; Insulin glulisine; Alzheimer's disease; Mild Cognitive Impairment; Intranasal insulin; Cognition Disorders
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Cognition Disorders | interventions — insulin glulisine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Insulin Glulisine (Experimental): Insulin Glulisine 20 IU (0.1ml/10 units in each nostril) per intranasal dose, 2 times per day for 6 months
  Interventions: Drug: Insulin glulisine
- Placebo (Placebo Comparator): Saline 20 IU (0.1 ml in each nostril) per intranasal dose, 2 times per day for 6 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Insulin glulisine
  Other Names: Apidra
  Arms: Insulin Glulisine
Drug: Placebo — Bacteriostatic 0.9% Sodium Chloride
  Other Names: Saline
  Arms: Placebo

SUMMARY:
This study evaluates the safety and effectiveness of intranasal (IN) glulisine in patients with amnestic mild cognitive impairment (aMCI) and probable Alzheimer's disease. Half of participants will receive IN glulisine, while the other half will receive IN placebo.

DETAILED DESCRIPTION:
Disruption of central nervous system (CNS) insulin signaling has been increasingly associated with Alzheimer's Disease pathogenesis, and consequently this disease has been referred to as a type III diabetes of the brain. Clinical trials of intranasal insulin in AD have demonstrated therapeutic effects of intranasal (IN) insulin in memory-impaired adults in terms of memory recall without significantly altering serum insulin or glucose levels. In this study, the investigators are investigating the chronic effects of the rapid acting insulin, glulisine, administered intranasally (IN) 20 IU two times daily in adults with amnestic-mild cognitive impairment (a-MCI) and mild Alzheimer's disease (AD). The investigation will enroll n=90 subjects and follow them over a 6 month period.

This study has the following objectives:

1. Primary:

   a. To measure the chronic effects of IN insulin glulisine on cognition and function in subjects with aMCI and probable mild AD over a 6 month period.
2. Secondary:

   1. To measure the effect of IN insulin glulisine on mood in subjects with aMCI and mild AD over a 6 month period.
   2. To measure the safety and efficacy of IN glulisine in aMCI and mild AD subjects with non-insulin dependent diabetes over a 6 month period.
3. Exploratory:

   1. To measure the effect of IN delivery of insulin glulisine on parieto-temporal and posterior cingulate/precuneus glucose metabolism in subjects with aMCI and mild AD over a 6 month period.
   2. To measure the chronic effect of IN delivery of insulin glulisine on AD-specific cerebrospinal (CSF) biomarkers (Abeta42, tau, and phospho-tau) in subjects with aMCI and mild AD over a 6 month period.

ELIGIBILITY:
Inclusion Criteria:

Subject is/has

* clinical and research diagnosis of amnestic-MCI OR probable mild AD in accordance with National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria
* Montreal Cognitive Assessment (MoCA) score 18-27
* Hachinski Ischemia Score <4
* 50-90 years of age
* Females at least 2 years post-menopausal or surgically sterile
* Proficiency in speaking, reading and understanding English
* Dedicated family member /caregiver, who will be able to attend all visits and report on subject's status
* (and family member/caregiver) provided fully informed written consent prior to participation. In the event that subject is legally unable to provide informed written consent due to deterioration in cognitive abilities, fully informed written consent must be provided by a legally authorized representative
* If AD, a brain computed tomography (CT) or magnetic resonance imaging (MRI) in the initial diagnostic workup or subsequent care that is compatible with the diagnosis of probable AD

Exclusion Criteria:

Subject has/have/is

* medical history and/or clinically determined evidence of other central nervous system (CNS) disorders including, but not limited to brain tumor, active subdural hematoma, seizure disorder, multiple sclerosis, dementia with Lewy bodies, vascular dementia, corticobasal syndrome, progressive supranuclear palsy, Parkinson's disease, multiple system atrophy, frontotemporal dementia, normal pressure hydrocephalus, Huntington's disease, or Jakob-Creutzfeldt disease presenting as dementia
* medical history and/or clinically determined disorders: current B12 deficiency, chronic sinusitis, any untreated thyroid disease, significant head trauma and history of difficulty with smell and/or taste prior to AD diagnosis
* history of any of the following: moderate to severe pulmonary disease, poorly controlled congestive heart failure, significant cardiovascular and/or cerebrovascular events within previous 6 months, condition known to affect absorption, distribution, metabolism, or excretion of drugs such as any hepatic, renal or gastrointestinal disease or any other clinically relevant abnormality that inclusion would pose a safety risk to the subject as determined by investigator
* previous nasal and/or oto-pharyngeal surgery and severe deviated septum and/or other anomalies
* history of any psychiatric illness, with the exception of major depressive and anxiety disorder (according to Diagnostic and Statistical Manual of Mental Disorders, version 5, Text Revision (DSM-IV TR)) currently in remission or stable with treatment for > 2 yrs, or any other psychiatric condition that inclusion would pose a safety risk to the subject as determined by investigator
* currently taking any medications, herbals and food supplements that are medically/clinically contraindicated as determined by investigator in order to comply with procedural testing of cognitive function as well as ensure study safety. See list of prohibited medications and compounds
* undergone a recent change (<1mo) in their prescribed acetylcholinesterase inhibitor (e.g. donepezil, rivastigmine, galantamine) or memantine.
* undergone a recent change (<1mo) in their selective serotonin re-uptake inhibitor (SSRI) or anti-depressant medication
* current or recent drug or alcohol abuse or dependence as defined by DSM-IV TR
* laboratory results that are medically relevant, in which inclusion would pose a safety risk to the subject as determined by investigator
* participated in any other research study at least 3 mos prior to this study
* an insulin allergy

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2015-09-28 (Actual); Primary Completion 2019-02-11 (Actual); Study Completion 2019-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Rosenbloom, MD, Principal Investigator — HealthPartners Institute
Locations (2):
- United States (2):
  - HealthPartners Riverside, Minneapolis, Minnesota
  - HealthPartners Neuroscience Center, Saint Paul, Minnesota

REFERENCES:
- [Derived] Rosenbloom M, Barclay TR, Kashyap B, Hage L, O'Keefe LR, Svitak A, Pyle M, Frey W, Hanson LR. A Phase II, Single-Center, Randomized, Double-Blind, Placebo-Controlled Study of the Safety and Therapeutic Efficacy of Intranasal Glulisine in Amnestic Mild Cognitive Impairment and Probable Mild Alzheimer's Disease. Drugs Aging. 2021 May;38(5):407-415. doi: 10.1007/s40266-021-00845-7. Epub 2021 Mar 15. PMID 33719017
- See also: HealthPartners Center for Memory and Aging — http://www.healthpartners.com/memoryloss

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 49 participants who signed a consent form for the study, 12 participants screen failed and did not meet the inclusion criteria at screening, 2 participants declined to participate after the initial screening. These 14 participants were not assigned to a treatment group since they were removed from the study prior to randomization.
Groups:
- Insulin Glulisine: Insulin Glulisine 20 IU (0.1ml/10 units in each nostril) per intranasal dose, 2 times per day for 6 months
  Insulin glulisine
Period: Overall Study
Arm/Group | Insulin Glulisine | Placebo
Started | 19 | 16
Completed | 18 | 13
Not Completed | 1 | 3
Not completed — Physician Decision | 1 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Insulin Glulisine | Placebo | Total
Number analyzed (Participants) | 19 | 16 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.4 (8.1) | 74.4 (6.4) | 71.1 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 10 | 10 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 19 | 16 | 35
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 18 | 12 | 30
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 19 | 16 | 35
Non-insulin dependent diabetes [Count of Participants; unit: Participants] | 3 | 2 | 5
Montreal cognitive assessment (MoCA) [Mean (Standard Deviation); unit: score on a scale] — The Montreal Cognitive Assessment (MoCA) was designed as a rapid screening instrument for mild cognitive dysfunction. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. The time to administer the MoCA is approximately 10 minutes. The scale ranges from 0-30 points, and scores of 26 or above are considered normal.
  score on a scale | 20.7 (2.1) | 21.1 (2.5) | 20.9 (2.3)
Diagnosis of probable mild Alzheimer's disease (AD) or amnestic mild cognitive impairment (aMCI) [Count of Participants; unit: Participants] — Diagnosis of AD or aMCI by a neurologist. aMCI is characterized by memory complaints and neuropsychological testing demonstrating abnormalities >1.0 standard deviation affecting memory with preservation of instrumental activities of daily living without functional limitations. The population has a 40% change of developing AD within 2 years. AD is chronic progressive neurodegenerative condition resulting in memory impairment, loss of function, and progressive deterioration in other cognitive domains like language, perceptual skills, attention, construction, orientation, and problem solving
  Participants
    Probable Mild AD | 10 | 11 | 21
    aMCI | 9 | 5 | 14
Apolipoprotein E4 (APOEe) status [Count of Participants; unit: Participants]
  Positive | 14 | 10 | 24
  Negative | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Change in Cognition as Measured by the Alzheimer's Disease Assessment Scale - Cognitive 13 (ADAS-Cog 13)
Description: The ADAS-Cog was developed as an outcome measure for global cognition in clinical trials for Alzheimer's disease. The ADAS-Cog assesses multiple cognitive domains including memory, language, praxis, and orientation. The modified ADAS-Cog 13-item scale includes all original ADAS-Cog items with the addition of a number cancellation task and a delayed free recall task, for a total of 85 points (0: no cognitive impairment; 85: severe impairment).
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Insulin Glulisine | Placebo
Number analyzed (Participants) | 16 | 12
score on a scale | 1.56 (4.2) | 0.81 (4.8)

2. Primary Outcome: Change in Functional Performance as Measured by the Clinical Dementia Rating (CDR) Scale
Description: The CDR is a 5-point scale used to characterize six domains of cognitive and functional performance applicable to Alzheimer disease and related dementias: Memory, Orientation, Judgment & Problem Solving, Community Affairs, Home & Hobbies, and Personal Care. Possible scores on the CDR are 0 (no impairment), 0.5 (very mild), 1 (mild), 2 (moderate), and 3 (severe). The total CDR ratings for each of the six cognitive/functional domains can be added to create a CDR sum of boxes (SOB). The overall SOB score ranges from 0 to 18; with 18 indicating severe impairment and 0 indicating no impairment.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Insulin Glulisine | Placebo
Number analyzed (Participants) | 16 | 12
score on a scale | 0.53 (.9) | -0.08 (1.5)

3. Primary Outcome: Change in Functional Performance as Measured by the Functional Activities Questionnaire (FAQ)
Description: The FAQ measures instrumental activities of daily living (IADLs), such as preparing balanced meals and managing personal finances. The FAQ is a sum of scores ranging from 0 (normal) to 30 (complete dependence on others).
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Insulin Glulisine | Placebo
Number analyzed (Participants) | 16 | 12
score on a scale | 2.5 (3.2) | 0.92 (3.4)

ADVERSE EVENTS:
Time Frame: 8 months
Description: Adverse event information was collected only from participants who were randomized to one of the two treatment groups. Participants who screen failed, withdrew, or were withdrawn prior to randomization are not included.
Arm/Group | Insulin Glulisine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/12
Serious Adverse Events (participants affected / at risk) | 1/16 | 0/12
Other Adverse Events (participants affected / at risk) | 17/19 | 10/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Glulisine (N=16) | Placebo (N=12)
Hospitalization (Renal and urinary disorders) | 1 (1) | 0 (0) — Dizziness secondary to dehydration and hyponatremia secondary to vomiting + hydrochlorothiazide
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Glulisine (N=19) | Placebo (N=16)
Nasal Irritation (Skin and subcutaneous tissue disorders) | 11 (11) | 5 (5)
Respiratory/Sinus symptoms (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 3 (3)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 3 (4) | 5 (8)
Imbalance/falls (General disorders) | 4 (4) | 3 (5)
Injury related to falls (General disorders) | 0 (0) | 3 (7)
Dental (Surgical and medical procedures) | 2 (3) | 1 (1)
Cardiovascular (Cardiac disorders) | 2 (2) | 2 (2)
Gastrointestinal (Gastrointestinal disorders) | 2 (4) | 2 (2)
Infection (Infections and infestations) | 2 (2) | 0 (0)
Nausea (General disorders) | 1 (1) | 1 (1)
Cancer (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Opthalmic (Eye disorders) | 1 (1) | 1 (1)
Hypoglycemia (General disorders) | 1 (1) | 0 (0)
Hematologic (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hearing Loss (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Endocrine (Endocrine disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-11): https://cdn.clinicaltrials.gov/large-docs/01/NCT02503501/Prot_SAP_001.pdf